CLINICAL TRIAL: NCT04877119
Title: Predictive Value for Preeclampsia of the sFlt-1:PlGF (Soluble Foms-like Tyrosine Kinase 1/Placental Growth Factor) Ratio in Pregnancy Complicated by Gestational Diabetes: The PREDICTION (PREeclampsia in DIabetiC gestaTION) Study
Brief Title: sFlt-1:PlGF Ratio in Gestational Diabetes: PREDICTION (PREeclampsia in DIabetiC gestaTION) Study
Acronym: PREDICTION
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Principal Investigator, Cristina Bianchi, Principal Investigator, Azienda Ospedaliero, Universitaria Pisana
Other Study IDs: 14905
Record Dates: First submitted 2021-04-29; First posted 2021-05-07 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Gestational Diabetes; Gestational Hypertension; Pre-Eclampsia
MeSH Terms: conditions — Diabetes, Gestational; Hypertension, Pregnancy-Induced; Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 25 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The ratio of soluble fms-like tyrosine kinase 1 (sFlt-1) to placental growth factor (PlGF) is elevated in pregnant women before the clinical onset of preeclampsia and can be used to predict the preeclampsia. However, its predictive value in pregnancy complicated by gestational diabetes is unclear. This study purposes are to validate a ratio of serum sFlt-1 to PlGF that would be predictive of the absence or presence of preeclampsia in the short term in women with singleton pregnancies complicated by diabetes in whom preeclampsia was suspected, and to evaluate the relationship among sFlt-1 to PlGF and placental histopathological alterations.

DETAILED DESCRIPTION:
Single center, observational, prospective study designed to validate a cutoff point of the sFlt-1:PlGF ratio for the prediction of the short-term absence or presence of preeclampsia in pregnancy complicated by gestational diabetes (GDM).

GDM women will be recruited at diabetes screening time (16-18 or 24-27 gestational weeks), performed according with the Italian National Guidelines by 75g - 2 hour Oral Glucose Tolerance Test. GDM will be defined according with International Association of Diabetes and Pregnancy Study Groups/World Health Organization 2013 criteria. A standardized medical history will be obtained in all the women at the time of their first visit, collecting data about maternal age, parity, last menstruation, pre-gestational weight, history of GDM, hypertension and macrosomia in previous pregnancies, family history of diabetes mellitus, education and employment. Moreover, during their visit, the women's weights were taken and their blood pressure measured. Blood samples for assessments of sFlt-1:PlGF ratio will be collected at visit 1 (baseline visit) and every 30±7 days after the previous visit until 36 gestational week (for a maximum of 4 determinations). At baseline and at each follow-up visits update of medical history, clinical assessments, laboratory testing and pregnancy evolution will be evaluated. During pregnancy all women will be receive standard diabetes and obstetric care, according with national guidelines. Diagnostic criteria for preeclampsia will be a new onset of both hypertension (systolic blood pressure ≥140 mmHg, diastolic blood pressure ≥90 mmHg, or both) and proteinuria (2+ protein or greater on dipstick urinalysis, ≥300 mg of protein per 24-hour urine collection, ≥30 mg /dl of protein in a spot urine sample, or a ratio of protein to creatinine of ≥30 mg/mmol) after 20 weeks of gestation. Only cases that met these prespecified criteria will be included in the analyses. At delivery, data items on maternal body weight at the end of pregnancy, time and mode of delivery, newborn bodyweight, preeclampsia as well as other maternal and fetal outcomes will be collected. Placental histopathological alterations will be detected in women who delivery by planned Cesarian section.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Diagnosis of GDM in the current pregnancy

Exclusion Criteria:

* Twin pregnancies
* Pre-pregnancy diabetes (type 1 or type 2 diabetes)
* Gestosis already diagnosed during the current pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Pregnant women with gestational diabetes
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-10-14 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Predictive SFLT-1 / PLGF ratio cat-off point for preeclampsia | 25 weeks
  Evaluation of a specific SFLT-1 / PLGF ratio cat-off point for women with diabetes during pregnancy (pre-pregnancy or gestational) in the prediction of preeclampsia

SECONDARY OUTCOMES:
Correlation between SFLT-1 / PLGF ratio and placental histopathology | 25 weeks
  Correlation between SFLT-1 / PLGF ratio and rate of placental histopathological alterations in pregnancy complicated by diabetes (pre-pregnancy or gestational)

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero-Universitaria Pisana - U.O. Malattie Metaboliche e Diabetologia, Pisa, PI, Italy

IPD SHARING:
Plan to Share IPD: No